CLINICAL TRIAL: NCT00177671
Title: Maintenance Therapies in Late-Life Depression: MTLD III
Brief Title: Antidepressant Medication Plus Donepezil for Treating Late-life Depression
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: R01MH043832-03 (NIH); R01MH043832 (NIH); 0312018; DATR A4-GPS
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2011-06-08 (Estimated); Last update posted 2013-02-06 (Estimated); Status verified 2013-01

CONDITIONS: Depression; Dementia
Keywords: Depression; Dementia; Alzheimer's Disease; Cognitive; Donepezil; Memory; Function; Elderly; Late-Life
MeSH Terms: conditions — Depression; Dementia; Alzheimer Disease | interventions — Escitalopram; Donepezil; Venlafaxine Hydrochloride; Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): escitalopram plus donepezil (DNP)in the experimental maintenance phase of the study.
  For subjects failing to respond to escitalopram during the initial open phase of acute treatment we allowed the use of duloxetine or venlafaxine to bring about remission and establish eligibility for randomized assignment to maintenance treatment with augmentation donepezil.
  Participants remained on the same antidepressant medication and dosage throughout the 2 year maintenance phase of the study. In the event of a recurrence of major depression during maintenance treatment, dosages of antidepressant medication were raised, or the antidepressant was switched to venlafaxine or duloxetine.
  For subjects failing to respond to escitalopram during the initial open phase of acute treatment, we allowed the use of duloxetine to bring about remission and establish eligibility for randomized assignment to maintenance treatment with augmentation placebo.
  Interventions: Drug: Escitalopram; Drug: Donepezil; Drug: Venlafaxine; Drug: Duloxetine
- 2 (Placebo Comparator): escitalopram plus placebo (PBO) in the experimental maintenance phase of the study.
  For subjects failing to respond to escitalopram during the initial open phase of acute treatment, we allowed the use of duloxetine or venlafaxine to bring about remission and establish eligibility for randomized assignment to maintenance treatment with augmentation placebo.
  Participants remained on the same antidepressant medication and dosage throughout the 2 year maintenance phase of the study. In the event of a recurrence of major depression during maintenance treatment, dosages of antidepressant medication were raised, or the antidepressant was switched to venlafaxine or duloxetine.
  For subjects failing to respond to escitalopram during the initial open phase of acute treatment, we allowed the use of venlafaxine or duloxetine to bring about remission and establish eligibility for randomized assignment to maintenance treatment with augmentation placebo.
  Interventions: Drug: Escitalopram; Drug: Venlafaxine; Drug: Placebo; Drug: Duloxetine

INTERVENTIONS:
Drug: Escitalopram — Escitalopram, 10mg to 20mg daily.
  Other Names: Lexapro
Drug: Donepezil — Donepezil, 5mg to 10mg daily.
  Other Names: aricept
  Arms: 1
Drug: Venlafaxine — Venlafaxine, 150mg to 300mg daily.
  Other Names: effexor XR
Drug: Placebo
  Arms: 2
Drug: Duloxetine
  Other Names: cymbalta

SUMMARY:
This study will determine the effectiveness of combining escitalopram, venlafaxine, or duloxetine with donepezil, a medication used in Alzheimer's disease, in improving memory, concentration, attention, and problem solving abilities, and reducing the risk of depressive relapse in older individuals with depression.

DETAILED DESCRIPTION:
The purpose of this research study is to learn if combining an antidepressant medication (escitalopram, venlafaxine, or duloxetine) with a medication used in Alzheimer's Disease (donepezil), in elderly patients age 65 and older with major depression, will help to 1) improve and/or maintain memory, concentration, attention, and problem solving abilities such as ability to balance a checkbook, pay bills, use the telephone, and 2) reduce the risk of depressive symptoms from returning. Study participation will last up to two years.

We aim to investigate pharmacologic strategies for improving and stabilizing cognitive functioning in late-life depression and minimizing progression of cognitive and associated functional impairment. Cognitive impairment in late-life depression has not been adequately addressed in previous intervention research, is a core feature of the illness, contributes markedly to disability and impaired quality of life, and is an overlooked but potentially critical target of intervention. Data from the MTLD II study suggest that treating depression does not normalize cognitive functions and may not prevent their progression. We will test a pharmacologic strategy involving the cholinesterase inhibitor donepezil, in combination with maintenance antidepressant pharmacotherapy (escitalopram, venlafaxine, or duloxetine), to improve and to maintain cognitive functioning and functional competence in elderly patients with major depression.

We hypothesize that maintenance antidepressant pharmacotherapy combined with donepezil will be superior to maintenance antidepressant pharmacotherapy combined with placebo/clinical management in (1) improving cognitive performance; and (2) slowing progression of cognitive impairment and decline in functional competence. We plan to recruit 200 patients aged 65 and above in current episodes of major depression. Those who respond to antidepressant pharmacotherapy with citalopram, venlafaxine, or duloxetine will then be randomly assigned on a double-blind basis to one of two 24-month treatments: 1)antidepressant pharmacotherapy plus donepezil/clinical management; or 2)antidepressant pharmacotherapy plus placebo/clinical management.

For information on related studies, please follow these links:

http://clinicaltrials.gov/show/NCT00000377

http://clinicaltrials.gov/show/NCT00178100

ELIGIBILITY:
Inclusion Criteria:

* Current episode of major depression
* HRS-D 17-item score of 15 or higher
* Must be able to speak English
* Willing to discontinue other psychotropics
* Availability of family member/caregiver
* Hearing capacity adequate to respond to raised conversational voice
* Must have no formal diagnosis of dementia

Exclusion Criteria:

* Meets DSM-IV criteria for bipolar disorder, schizophrenia, schizoaffective disorder, or a psychotic disorders
* Alcohol/drug abuse within 12 months of study entry
* History of treatment non-adherence in other clinic protocols
* History of non-response to citalopram in other clinic protocols
* History of non-tolerance to SSRI therapy

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 220 (Actual)
Dates: Start 2003-12; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bruce G. Pollock, MD, PhD, Principal Investigator — University of Pittsburgh Professor of Psychiatry, Pharmacology, and Nursing
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Reynolds CF 3rd, Butters MA, Lopez O, Pollock BG, Dew MA, Mulsant BH, Lenze EJ, Holm M, Rogers JC, Mazumdar S, Houck PR, Begley A, Anderson S, Karp JF, Miller MD, Whyte EM, Stack J, Gildengers A, Szanto K, Bensasi S, Kaufer DI, Kamboh MI, DeKosky ST. Maintenance treatment of depression in old age: a randomized, double-blind, placebo-controlled evaluation of the efficacy and safety of donepezil combined with antidepressant pharmacotherapy. Arch Gen Psychiatry. 2011 Jan;68(1):51-60. doi: 10.1001/archgenpsychiatry.2010.184. PMID 21199965
- [Derived] Diniz BS, Reynolds CF 3rd, Begley A, Dew MA, Anderson SJ, Lotrich F, Erickson KI, Lopez O, Aizenstein H, Sibille EL, Butters MA. Brain-derived neurotrophic factor levels in late-life depression and comorbid mild cognitive impairment: a longitudinal study. J Psychiatr Res. 2014 Feb;49:96-101. doi: 10.1016/j.jpsychires.2013.11.004. Epub 2013 Nov 20. PMID 24290367
- [Derived] Andreescu C, Tudorascu DL, Butters MA, Tamburo E, Patel M, Price J, Karp JF, Reynolds CF 3rd, Aizenstein H. Resting state functional connectivity and treatment response in late-life depression. Psychiatry Res. 2013 Dec 30;214(3):313-21. doi: 10.1016/j.pscychresns.2013.08.007. Epub 2013 Oct 18. PMID 24144505
- [Derived] Sheffrin M, Driscoll HC, Lenze EJ, Mulsant BH, Pollock BG, Miller MD, Butters MA, Dew MA, Reynolds CF 3rd. Pilot study of augmentation with aripiprazole for incomplete response in late-life depression: getting to remission. J Clin Psychiatry. 2009 Feb;70(2):208-13. doi: 10.4088/jcp.07m03805. Epub 2009 Feb 10. PMID 19210951
- [Derived] Karp JF, Whyte EM, Lenze EJ, Dew MA, Begley A, Miller MD, Reynolds CF 3rd. Rescue pharmacotherapy with duloxetine for selective serotonin reuptake inhibitor nonresponders in late-life depression: outcome and tolerability. J Clin Psychiatry. 2008 Mar;69(3):457-63. doi: 10.4088/jcp.v69n0317. PMID 18251622

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 220 signed consent; 158 participants completed pre-randomization testing; 130 participants were randomized. Of these 130, 67 randomized to donepezil augmentation and 63 to placebo.
Pre-assignment Details: 28 enrolled participants were not randomized due to the following reasons: dementia (19), consent withdrawal (4), con-compliance with research procedures (3), supervening medical problems that precluded participation (2).
Groups:
- Donepezil: Treatment with antidepressants (escitalopram (10mg to 20mg daily), venlafaxine (150mg to 300mg daily), duloxetine(20mg to 120mg daily) plus donepezil (5mg to 10mg daily)
- Placebo: Treatment with antidepressants (escitalopram (10mg to 20mg daily), venlafaxine (150mg to 300mg daily), duloxetine(20mg to 120mg daily) plus placebo
Period: Overall Study
Arm/Group | Donepezil | Placebo
Started | 67 | 63
Month 12 | 45 | 57
Month 24 | 42 | 49
Completed | 42 | 49
Not Completed | 25 | 14
Not completed — Withdrawal by Subject | 5 | 6
Not completed — medical complications | 2 | 0
Not completed — Adverse Event | 6 | 0
Not completed — Physician Decision | 12 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Donepezil | Placebo | Total
Number analyzed (Participants) | 67 | 63 | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 67 | 63 | 130
Age Continuous [Mean (Standard Deviation); unit: years] | 73.1 (6.5) | 73.9 (5.8) | 73.5 (6.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 51 | 100
  Male | 18 | 12 | 30
Region of Enrollment [Number; unit: participants]
  United States | 67 | 63 | 130

OUTCOME MEASURES:

1. Primary Outcome: Global Cognitive Performance
Description: Cognitive performance was assessed with 17 well established and validated individual tests measuring multiple domains. We transformed raw scores for individual tests into Z-scores using the baseline distribution of a non-depressed, cognitively normal, older adult comparison group (N=36)of similar age, education, and medical health recruited concurrently with the depressed participants. These Z-scores were averaged within each neuropsychological area to produce domain scores and then averaged over all 17 tests to calculate a global cognition performance score.
Time Frame: Measured at baseline and Years 1 and 2 in maintenance
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 67 | 63
Z-score
  Baseline (N=67;N=63) | -0.47 (0.88) | -0.47 (0.76)
  Year 1 (N=45; N=57) | -0.23 (0.79) | -0.65 (0.81)
  Year 2 N=42; N=49) | -0.31 (0.92) | -0.56 (0.90)

2. Primary Outcome: Cognitive Instrumental Activities of Daily Living (IADL)
Description: The PASS (a performance-based assessment of instrumental activities of daily living)generates a composite measure of 13 cognitive IADL items capturing performance on activities such as shopping, bill paying, medication management, and home safety. We report the percentage of subjects at each assessment point adjudged to have independent functioning. This was determined by a clinician rater observing subjects perform each task and rating them according to predetermined criteria on a 4 point scale, ranging from 0 (unable) to 3 (independent).
Time Frame: baseline, year 1 and year 2
Population: Some participants refused this testing.
Measure: Number; unit: Percentage of participants
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 33 | 34
Percentage of participants
  Baseline (N=33; N=34) | 54.10 | 61.82
  Year 1 (N=23; N=25) | 62.16 | 54.35
  Year 2 (N=11; N=17) | 36.67 | 47.22

3. Primary Outcome: Number of Participants With Recurrence of Major Depression
Description: Recurrence of major depressive episodes as determined by SCID/DSM IV: two weeks of low mood and/or anhedonia, together with at least five of the following symptoms: suicidal ideation, low energy, sleep disturbance, appetite disturbance, psychic anxiety or somatic anxiety. In addition, a diagnosis of major depression requires evidence of distress or impairment.
Time Frame: 2 years
Measure: Number (95% Confidence Interval); unit: participants
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 67 | 63
participants | 19 [16 to 31] | 11 [6 to 18]
Statistical Analysis 1: Comparison: Donepezil vs Placebo; We followed the intention to treat principle. We used Kaplan-Meier curves to quantify the percentage of participants who were free of depression recurrence over time. Cox proportional hazard models quantified hazard ratios comparing the 2 treatment groups; Test type: Superiority or Other; p = .05, Log Rank; Hazard Ratio (HR) = 3.97, 95% CI 2-sided [1.00 to 4.41], Standard Deviation 2.09

4. Post Hoc Outcome: Percentage of Participants With Mild Cognitive Impairment Converting to Dementia.
Description: Conversion to dementia was ascertained by the University of Pittsburgh Alzheimer Disease Research Center (ADRC), using data on neuropsychological performance and IADL functioning, as well as other relevant clinical data. Diagnoses were made according to National Alzheimer Coordinating Center criteria.
Time Frame: 2 year
Population: This is the percent of participants with mild cognitive impairment (MCI) in each arm of the study.
Measure: Number; unit: Percent of Participants
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 30 | 27
Percent of Participants | 10 | 33

ADVERSE EVENTS:
Time Frame: 2 years
Description: We determined adverse events by structured clinical interview.
Arm/Group | Donepezil | Placebo
Serious Adverse Events (participants affected / at risk) | 3/67 | 1/63
Other Adverse Events (participants affected / at risk) | 0/67 | 0/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=67) | Placebo (N=63)
Suicide Attempt (Psychiatric disorders) | 1 (1) | 0 (0)
stroke (Nervous system disorders) | 1 (1) | 0 (0)
Myocardial infarcation with congestive heart failure (Cardiac disorders) | 1 (1) | 0 (0)
Death due to heart attack in person with history of coronary heart disease and hypertension. (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Observations about dementia conversion rates were obtained from post hoc subgroup analyses of participants with mild cognitive impairment (N=57) and participants with normal cognition at time of randomization (N=63).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No